CLINICAL TRIAL: NCT00270140
Title: A Double-Blind, Placebo-Controlled Study to Determine the Safety and Efficacy of Multiple Doses of R-HuEPO in Facilitating Presurgical Autologous Blood Donation
Brief Title: A Study to Evaluate the Safety and Effectiveness of Epoetin Alfa Versus Placebo in Facilitating the Presurgical Collection of Blood to be Used for Self-donation During Surgery on the Spine, Hip, or Knee.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005920
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-02

CONDITIONS: Anemia; Blood Transfusions, Autologous; Orthopedic Procedures
Keywords: anemia; blood transfusion; epoetin alfa; erythropoietin; surgery; blood donation; blood
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa at doses of 150, 300, or 600 units per kilogram of body weight versus placebo in facilitating presurgical collection of blood for self-donation during surgery of the knee, hip or spine. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Major surgical procedures may require transfusion of several units of blood. Blood transfusions from other people may be associated with transfusion reactions that cause fever or with viral infections that can be carried (and donated) in blood. However, self-donations of blood may cause anemia in a patient who will be undergoing surgery a few weeks later. Previous research with epoetin alfa suggests that epoetin alfa speeds up the rate of red blood cell production and has a beneficial effect on anemia. This randomized, double-blind, placebo-controlled, multicenter study is designed to determine whether treating patients with epoetin alfa will stimulate a person's bone marrow to produce red blood cells and therefore increase a patient's ability to self-donate blood prior to major surgery for joint diseases. Patients will be randomly assigned to receive 150, 300, or 600 units of epoetin alfa per kilogram of body weight, or matching placebo, injected into a vein on the first study day, and every 3 to 4 days thereafter for 21 days. Effectiveness will be determined by the number of units of blood that can be donated by patients during the study, the number of units of non-self-donated blood used during surgery, the total red cell volume of the self-donated blood, the total red cell production, and the percentage of sub-standard units of blood that are self-donated. Safety evaluations including the incidence of adverse events, physical examinations, and clinical laboratory tests will be performed throughout the study. The study hypothesis is that patients treated with epoetin alfa will be able to donate more units of blood than those patients who receive placebo. Epoetin alfa, 150, 300, or 600 units per kilogram of body weight, or placebo, injected into a vein every three to four days for 21 days (6 doses) during the period before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery on the knee, hip, or spine between 25 and 35 days after starting epoetin alfa therapy
* having a hematocrit (percentage of red cells in the blood) of >39 percent and <=50 percent
* in good general health

Exclusion Criteria:

* Patients having a history of any primary blood disease
* having a history of artery blockage in the heart, body or brain, or a history of seizures
* having uncontrolled high blood pressure, a folate deficiency, vitamin B12 deficiency or iron deficiency anemia, active inflammatory disease (except osteoarthritis or rheumatoid arthritis) or a disease that destroys blood cells
* losing blood from the stomach, intestines or elsewhere in the body
* having received therapy with any drug known to affect red blood cell formation (such as chemotherapy for cancer)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1989-09; Study Completion 1991-08 (Actual)

PRIMARY OUTCOMES:
Number of units of units of blood donated by the patient; Number of units of donor blood transfused during surgery; Total red cell volume and percentage in self-donated blood; Percentage of sub-standard units of blood self-donated

SECONDARY OUTCOMES:
Percentage in each treatment group of patients requiring blood donated by others; Safety evaluations including the incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the safety and effectiveness of epoetin alfa in facilitating the presurgical collection of blood to be used for self-donation during surgery on the spine, hip, or knee. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=685&filename=CR005920_CSR.pdf